CLINICAL TRIAL: NCT04189042
Title: Assessing Validity and Reliability of Figure-of-Eight Walk Test in People With Parkinson's Disease
Brief Title: Figure-of-Eight Walk Test in Parkinson
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Çağrı Gülşen, Principal Investigator, Gazi University
Other Study IDs: 2019.19.164
Record Dates: First submitted 2019-12-04; First posted 2019-12-06 (Actual); Last update posted 2021-02-04 (Actual); Status verified 2021-02

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Week
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Parkinson Group: Patients with Parkinson's Disease (Hoehn and Yahr stage 1-4)
- Healthy Control: Healthy People

SUMMARY:
The aim of study is to assess validity and reliability of Figure-of-Eight Walk Test in people with Parkinson's Disease

ELIGIBILITY:
Inclusion Criteria:

* at least 40 years of age
* neurologist-diagnosed Parkinson's Disease
* Hoehn & Yahr (H&Y) stages 1 to 3
* able to walk at least 20 meters

Exclusion Criteria:

* other neurologic disorder
* visual, auditory, orientational problems that could affect study results
* any orthopedic problem that prevents walking and standing
* have a cardiovascular, pulmonary or hormonal disorder

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with Parkinson's Disease who apply to the Gazi University, Department of Physiotherapy and Rehabilitation will be invited to this study.
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2019-12-11 (Actual); Primary Completion 2021-03-30 (Estimated); Study Completion 2021-05-31 (Estimated)

PRIMARY OUTCOMES:
Figure-of-Eight Walk Test | 10-15 seconds
  Figure-of-Eight Walk Test involves straight and curved paths in order to assess the advanced walking performance required in daily life.The subject walks a "figure 8" pattern around two cones spaced 5 ft apart, and the time and number of steps needed to complete the assessment are recorded.

SECONDARY OUTCOMES:
Unified Parkinson's Disease Rating Scale | 15 minutes
  The Unified Parkinson's Disease Rating Scale (UPDRS) is a widely used measure of impairment and disability associated with Parkinson's Disease (PD) consisting of four sections: (1) Mentation, behavior, and mood; (2) Activities of daily living (ADLs); (3) Motor; and (4) Complications.Sections I through III are scored using a 5-point Likert-type scale (0 = no impairment; 4 = marked impairment). Although individual sections are scored and reported independently, scores from sections I through III are also summed to provide a UPDRS Total score. The UPDRS total score ranges between 0 and 199 points. Higher points indicates worse outcome.
Hoehn and Yahr Scale | 1 minutes
  Disease stage is assessed by the Hoehn and Yahr Scale. The Hoehn and Yahr scale is a commonly used diagnostic tool for quantifying the progression of Parkinson's Disease symptoms. Stages range from 0 (no signs of disease) to 5 (requiring a wheelchair, or bedridden unless assisted).
Timed Up and Go Test | 10-15 seconds
  Functional mobility is assessed by using the timed up and go test. The timed up and go test measures the time that a patient needs to stand up from a chair, walk a 3-m distance, come back and sit back on the chair.
Berg Balance Scale | 10-15 minutes
  Berg Balance Scale (BBS) is a scale that using for assess postural stability. It ranges 0-56 with higher score indicates better stability.
10 Meter Walk Test | 10-15 seconds
  10 Meter Walk Test measures the time required to complete straight walk of 10 meters distance.
Activities-Specific Balance Confidence (ABC) Scale | 5 minutes
  Activities-specific Balance Confidence scale (ABC), to quantify the level of confidence in performing a specific task without losing balance or becoming unsteady.The ABC scale is a self-reported questionnaire providing information on balance confidence in the performance of 16 different daily activities, such as stair climbing, walking in the house, and walking on slippery floors. The questionnaire contains 16 items scored on a range from 0% to 100% (0 indicating no confidence and 100 indicating full confidence).

CONTACTS AND LOCATIONS:
Locations (1):
- Gazi University, Faculty of Health Sciences, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No